CLINICAL TRIAL: NCT00736320
Title: HD16 for Early Stages - Treatment Optimization Trial in the First-line Treatment of Early Stage Hodgkin Lymphoma; Treatment Stratification by Means of FDG-PET
Brief Title: HD16 for Early Stage Hodgkin Lymphoma
Acronym: HD16
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD16
Record Dates: First submitted 2008-08-08; First posted 2008-08-15 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; early stage; PET
MeSH Terms: conditions — Hodgkin Disease | interventions — ABVD protocol; Doxorubicin; Bleomycin; Vincristine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 2 cycles ABVD followed by 20 Gy IF-RT irrespective of FDG-PET results after chemotherapy
  Interventions: Drug: ABVD (Adriamycin, Bleomycin, Vincristine, Dacarbazine); Radiation: 20 Gy IFRT (Involved Field Radiotherapy)
- B (Experimental): 2 cycles ABVD followed by 20 Gy IF-RT if FDG-PET is positive after chemotherapy; 2 cycles ABVD and treatment stop if FDG-PET is negative after chemotherapy
  Interventions: Drug: ABVD (Adriamycin, Bleomycin, Vincristine, Dacarbazine); Radiation: 20 Gy IFRT (Involved Field Radiotherapy)

INTERVENTIONS:
Drug: ABVD (Adriamycin, Bleomycin, Vincristine, Dacarbazine) — chemotherapy with 2 cycles of ABVD (day 1 + 15)
Radiation: 20 Gy IFRT (Involved Field Radiotherapy) — 20 Gy Involved Field Radiotherapy

SUMMARY:
This study is designed to test the non-inferiority of the experimental arm compared to the standard arm in terms of Progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin Lymphoma
* CS I, II without risk factors

  * large mediastinal mass (> 1/3 of maximum transverse thorax diameter)
  * extranodal involvement
  * elevated ESR
  * 3 or more involved nodal areas
* Written informed consent

Exclusion Criteria:

* Leucocytes < 3000/µl
* Platelets < 100000/µl
* Hodgkin Lymphoma as composite lymphoma
* Activity index (WHO) > 2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2009-11; Primary Completion 2018-09 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 5 years

SECONDARY OUTCOMES:
overall survival | 5 years
acute toxicity | 5 years
late toxicity | 5 years
CR rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University of Cologne
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- [Derived] Lommen M, Weindler JJ, Jablonski J, Rosenbrock J, Borchmann P, Behringer K, Roth KS, Ufton D, Dietlein M, Kobe C, Ferdinandus J. Association between metabolic tumor burden and health-related quality of life in patients with classic Hodgkin lymphoma. Eur J Nucl Med Mol Imaging. 2025 Oct 11. doi: 10.1007/s00259-025-07569-5. Online ahead of print. PMID 41074963
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] van Heek L, Stuka C, Kaul H, Muller H, Mettler J, Hitz F, Baues C, Fuchs M, Borchmann P, Engert A, Dietlein M, Voltin CA, Kobe C. Predictive value of baseline metabolic tumor volume in early-stage favorable Hodgkin Lymphoma - Data from the prospective, multicenter phase III HD16 trial. BMC Cancer. 2022 Jun 18;22(1):672. doi: 10.1186/s12885-022-09758-z. PMID 35717166
- [Derived] Fuchs M, Goergen H, Kobe C, Kuhnert G, Lohri A, Greil R, Sasse S, Topp MS, Schafer E, Hertenstein B, Soekler M, Vogelhuber M, Zijlstra JM, Keller UB, Krause SW, Wilhelm M, Maschmeyer G, Thiemer J, Duhrsen U, Meissner J, Viardot A, Eich H, Baues C, Diehl V, Rosenwald A, von Tresckow B, Dietlein M, Borchmann P, Engert A. Positron Emission Tomography-Guided Treatment in Early-Stage Favorable Hodgkin Lymphoma: Final Results of the International, Randomized Phase III HD16 Trial by the German Hodgkin Study Group. J Clin Oncol. 2019 Nov 1;37(31):2835-2845. doi: 10.1200/JCO.19.00964. Epub 2019 Sep 10. PMID 31498753
- [Derived] Voltin CA, Goergen H, Baues C, Fuchs M, Mettler J, Kreissl S, Oertl J, Klaeser B, Moccia A, Drzezga A, Engert A, Borchmann P, Dietlein M, Kobe C. Value of bone marrow biopsy in Hodgkin lymphoma patients staged by FDG PET: results from the German Hodgkin Study Group trials HD16, HD17, and HD18. Ann Oncol. 2018 Sep 1;29(9):1926-1931. doi: 10.1093/annonc/mdy250. PMID 30010775
- [Derived] Narang AK, Terezakis SA. Contemporary radiation therapy in combined modality therapy for Hodgkin lymphoma. J Natl Compr Canc Netw. 2015 May;13(5):597-605. doi: 10.6004/jnccn.2015.0077. PMID 25964643
- See also: Homepage GHSG — http://www.ghsg.org